CLINICAL TRIAL: NCT01001338
Title: Randomized, Double-Blind, Multicenter, Placebo-Controlled, Combination Study to Evaluate the Safety, Efficacy and Potential Pharmacokinetic Interaction of RDEA594 and Allopurinol in Gout Patients With an Inadequate Hypouricemic Response With Standard Doses of Allopurinol
Brief Title: Allopurinol Combination Study
Acronym: RDEA594-203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: RDEA594-203
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- RDEA594 200 mg qd (Experimental): RDEA594 200 mg qd plus allopurinol qd
  Interventions: Drug: RDEA594; Drug: Allopurinol
- RDEA594 200 mg, 400 mg qd (Experimental): RDEA594 200 mg then 400 mg qd plus allopurinol qd.
  Patients on lesinurad 400 mg had their dose changed to lesinurad 200 mg after protocol amendment 16 dated 07 October 2015.
  Interventions: Drug: RDEA594; Drug: Allopurinol
- Matching Placebo (Placebo Comparator): RDEA594 matching placebo qd plus allopurinol qd, then allopurinol qd alone in open label period.
  Patients on allopurinol qd alone were discontinued after protocol amendment 16 dated 07 October 2015.
  Interventions: Drug: Placebo; Drug: Allopurinol
- RDEA594 600 mg qd (Experimental): RDEA594 200 mg then 400 mg then 600 mg plus allopurinol qd
  Patients on lesinurad 600 mg had their dose changed to lesinurad 200 mg after protocol amendment 16 dated 07 October 2015.
  Interventions: Drug: RDEA594; Drug: Allopurinol

INTERVENTIONS:
Drug: RDEA594 — Uricosuric agent for the treatment of gout.
  Arms: RDEA594 200 mg qd; RDEA594 200 mg, 400 mg qd; RDEA594 600 mg qd
Drug: Placebo — Matching Placebo
  Arms: Matching Placebo
Drug: Allopurinol — Allopurinol

SUMMARY:
To compare the proportion of subjects whose serum urate (sUA) levels are < 6.0 mg/dL following 4 weeks of continuous treatment of RDEA594 in combination with allopurinol to allopurinol alone in subjects with documented inadequate hypouricemic response with standard doses of allopurinol.

ELIGIBILITY:
Inclusion Criteria:

1. Male or a post-menopausal or surgically sterile female.
2. 18 - 80 years of age.
3. Has been taking allopurinol as the sole urate lowering therapy for hyperuricemia for at least 6 weeks at a dose between 200 mg and 600 mg per day without an adequate response.
4. Has a sUA level ≥ 6 mg/dL at screening.
5. Meets criteria for the diagnosis of gout as per the American Rheumatism Association (ARA) Criteria for the Classification of Acute Arthritis of Primary Gout.
6. Willing and able to give informed consent and adhere to visit/protocol schedules (informed consent must be given before the first study procedure is performed).
7. Subjects entering the optional Extension Period must have completed 28 days of dosing in the Double-Blind Treatment Period and the Day 42 Visit in the Follow-up Period within 4 months and must not have experienced any serious adverse events considered possibly related to study drug.
8. Subjects entering the optional Open-Label Extension Period must continue to be compliant with the protocol through Week 44 of the Double-Blind Extension Period and must not have experienced any serious adverse events considered possibly related to study drug.

Exclusion Criteria:

1. Consumes more than 14 drinks of alcohol per week (e.g., 1 drink = 5 oz [150 ml] of wine, 12 oz [360 ml] of beer, or 1.5 oz [45 ml] of hard liquor).
2. History or suspicion of drug abuse.
3. History of documented or suspected kidney stones.
4. Has rheumatoid arthritis or other autoimmune disease requiring treatment.
5. Documented or suspicion of HIV infection.
6. Positive serology to HCV antibodies (Abs), and/or hepatitis B surface antigen (HBsAg).
7. History of malignancy within 5 years prior to the first dose of study medication, other than non-melanomatous skin cancer or cervical dysplasia.
8. History of cardiac abnormalities, including abnormal and clinically relevant ECG changes
9. Any condition predisposing to QT prolongation including pathological Q-wave (defined as Q-wave >40 msec or depth > 0.4-0.5 mV).
10. Any use of concomitant medications that prolong the QT/QTc interval within the 14 days prior to Baseline (Day 1).
11. QT interval corrected for heart rate according to Fridericia (QTcF) > 450 msec at Screening or pre-dose at Baseline (Day 1).
12. Uncontrolled hypertension (above 150/95).
13. Inadequate renal function [serum creatinine >1.5 mg/dL or creatinine clearance < 60 mL/min (by Cockroft-Gault formula)].
14. Hemoglobin < 10 g/dL (males) or < 9 g/dL (females).
15. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN).
16. Gamma glutamyl transferase (GGT) > 3 x ULN.
17. Active peptic ulcer disease requiring treatment.
18. History of xanthinuria, active liver disease, or hepatic dysfunction.
19. Requires therapy with any other urate-lowering medication, other than the study medications.
20. Requires long-term use of salicylates; diuretics; losartan; azathioprine; mercaptopurine; theophylline; intravenous colchicine; cyclosporine; cyclophosphamide; pyrazinamide; sulfamethoxazole; or trimethoprim.
21. Taking medications known as enzyme inducers (see section 3.7 for listing).
22. Reports receiving a strong or moderate inhibitor of CYP3A4 or a P-gp inhibitor within 1 month prior to study drug dosing, due to potential interactions with colchicine.
23. Acute gout flare (exclusive of chronic synovitis/ arthritis) during the Screening-Period that has not resolved one week prior to the Baseline Visit (Day 0).
24. Pregnant or breast feeding.
25. Has received an investigational medication within 4 weeks prior to the screening visit for this study.
26. Previously participated in a clinical study involving RDEA806 or RDEA594.
27. Known hypersensitivity or allergy to RDEA594, allopurinol or colchicine or any components in their formulations.
28. Body mass index (BMI) >48 kg/m2.
29. Taking greater than 1000 mg/day of Vitamin C.
30. Any other medical or psychological condition, which in the opinion of the Investigator and/or Medical Monitor, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements, or to complete the study.
31. Inadequate renal function after completing the Double-Blind Treatment period prior to entering Double-Blind Extension Period.
32. Requiring treatment with prohibited medications noted in exclusion criteria numbers 20-23 after completing the Double-Blind Treatment Period prior to entering the Extension Period.
33. Clinically relevant medical event as determined by the investigator in consultation with medical monitor prior to entering the Extension Period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To compare the percent reduction from baseline in serum urate levels following 4 wks of continuous treatment of RDEA594 in combination with allopurinol to allopurinol alone in subjects with documented inadequate hypouricemic response. | 28 days

SECONDARY OUTCOMES:
To evaluate the proportion of subjects whose sUA levels are < 6.0 mg/dL, < 5.0 mg/dL and < 4.0 mg/dL at each study visit by treatment group in all subjects and in subjects who have an sUA ≥6 mg/dL at the baseline visit. | 28 days and through extension
To evaluate the absolute and percent reduction from baseline in sUA levels at each visit. | 28 days and through extension
To evaluate the percentage change in 24-hour urine urate level (excretion) from baseline to Day 28. | 28 days and through extension
To evaluate the incidence of gout flares. | 28 days and through extension
To evaluate the safety and tolerability of RDEA594 in combination with allopurinol in subjects with gout. | 28 days and through extension
To compare the multiple-dose pharmacokinetics (PK) of allopurinol and oxypurinol in the absence versus presence of RDEA594 co-administration. | 28 days
To evaluate the proportion of subjects whose sUA level decreases to or is maintained at <6.0 mg/dL and <5.0 mg/dL in the Double-Blind and Open-Label Extension Period. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nihar Bhakta, MD, Study Director — Ardea Biosciences, Inc.
Locations (43):
- United States (25):
  - Phoenix, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Stanford, California
  - Boca Raton, Florida
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Jupiter, Florida
  - Meridan, Idaho
  - Lexington, Kentucky
  - Wheaton, Maryland
  - Las Vegas, Nevada
  - Reno, Nevada
  - Harrisburg, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mayfield Village, Ohio
  - Durham, South Carolina
  - Rock Hill, South Carolina
  - Germantown, Tennessee
  - Jackson, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - West Jordan, Utah
  - Chesapeake, Virginia
- Canada (6):
  - Coquitlam, British Columbia
  - Kelowna, British Columbia
  - St. John's, Newfoundland and Labrador
  - Thornhill, Ontario
  - Toronto, Ontario
  - Mirabel, Quebec
- Poland (6):
  - Bydgoszcz
  - Elblag
  - Lublin
  - Poznan
  - Radom
  - Torun
- Bilbao, Spain
- Ukraine (4):
  - Donetsk
  - Kharkiv
  - Kyiv
  - Vinnytsia
- Blackpool, Lancashire, United Kingdom

REFERENCES:
- [Derived] Perez-Ruiz F, Sundy JS, Miner JN, Cravets M, Storgard C; RDEA594-203 Study Group. Lesinurad in combination with allopurinol: results of a phase 2, randomised, double-blind study in patients with gout with an inadequate response to allopurinol. Ann Rheum Dis. 2016 Jun;75(6):1074-80. doi: 10.1136/annrheumdis-2015-207919. Epub 2016 Jan 7. PMID 26742777